CLINICAL TRIAL: NCT04664920
Title: An Individualized Exergame Training Solution for People With Major Neurocognitive Disorder: a Usability Study
Status: Completed | Type: Observational
Sponsor: Davy Vancampfort (Other)
Responsible Party: Sponsor-Investigator, Davy Vancampfort, Professor, KU Leuven
Organization: KU Leuven (Other)
Other Study IDs: 052020
Record Dates: First submitted 2020-06-03; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Major Neurocognitive Disorder; Physical Activity; Dementia
MeSH Terms: conditions — Motor Activity; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Exergame intervention arm.
  Interventions: Device: exergame

INTERVENTIONS:
Device: exergame — motor-cognitive training device

SUMMARY:
The aim of this study is to investigate the usability of a newly designed and developed user-centered exergame in older adults with major neurocognitive disorder (dementia).

DETAILED DESCRIPTION:
The aim of this study is to investigate the usability of a newly designed and developed user-centered exergame in older adults with major neurocognitive disorder (dementia). On one appointment, the participants will perform a user-centered exergame for about 30 minutes. The exergame will include specific cognitive and motor functions. As the difficulty of the training game is user-centered, the participants will always be challenged on an appropriate level. Stepping exercises will be used to control the video game scenario. The video game scenario will include different cognitive functions. The body movements will include different physical aspects including balance, strength and Pelvic Floor Muscle Training (PFMT). During the exergame performance, different qualitative assessments will be performed to determine usability of the exergame including acceptance and game experience protocol (think aloud method). After the exergame performance, the participant will answer individual and guideline-based interview questions about usability including their individual experiences (duration about 20 min). This study contributes to fundamental research investigating how user-centered exergame training can be applied in older adults with individual needs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60+ years
* Live in long-term care facility "de Wingerd"
* Being diagnosed with major neurocognitive disorder by a specialist doctor
* Standing straight for minimal 10 minutes without aids
* Visual acuity with correction sufficient to work on a TV screen

Exclusion Criteria:

* Mobility impairments that don't allow to play the exergame
* Severe acute or uncontrolled health problems (e.g. recent cardiac infarction, uncontrolled diabetes or hypertension)
* Orthopaedic or neurological diseases that inhibit Exergame training
* Rapidly progressive or terminal illness

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Residents of long-term care facility 'de Wingerd'.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Acceptance questionnaire | 2 years
  users' individual acceptance
Game experience questionnaire | 2 years
  users' game experience
Guideline-based qualitative interview | 2 years
  Users' opinions and feedback
System usability questionnaire | 2 years
  System usability scale

CONTACTS AND LOCATIONS:
Locations (1):
- De Wingerd, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No